CLINICAL TRIAL: NCT03089424
Title: Effects of Photobiomodulation Therapy in Patients With Chronic Non-specific Low Back Pain: a Randomized Placebo-controlled Trial
Brief Title: Photobiomodulation Therapy on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Shaiane da Silva Tomazoni, Postdoctoral fellow, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.964.094
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain
Keywords: low back pain, photobiomodulation therapy, LLLT
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The mode of intervention (active or placebo photobiomodulation) will be coded by an independent researcher. The randomization schedule will contain only codes (not the actual intervention). The output from the laser device is exactly the same from either the active or the placebo interventions. These features will guarantee that participants, therapists and outcomes assessor will be blinded to the treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo PBMT (Placebo Comparator): Application of PBMT (Photobiomodulation Therapy) without any dose (0 Joule) and The Back Book (educational information booklet).
  Interventions: Device: Placebo PBMT
- PBMT active (Active Comparator): Application of PBMT (Photobiomodulation Therapy) active and The Back Book (educational information booklet).
  Interventions: Device: PBMT active

INTERVENTIONS:
Device: Placebo PBMT — The PBMT treatments will be performed using the Multi Radiance Medical™ Super Pulsed Laser MR4™ console (Solon, OH, USA), with the LS50 (emitter with an area of 20 cm2) and SE25 (emitter with an area of 4 cm2) cluster probes as emitters. Nine sites will be irradiated at patient's lumbar region: 3 central sites, using the SE25 (without any dose, 0 J); and 6 sites in the same direction, but laterally (both sides, 3 at a side), using the LS50 (without any dose, 0 J). Patients will be treated during 12 sessions over a period of four weeks (three sessions/week). At each treatment session, patients will receive a total dose of 0 J. At the end of the 12 treatment sessions, patients will receive a total dose of 0 J.
  Arms: Placebo PBMT
Device: PBMT active — The PBMT treatments will be performed using the Multi Radiance Medical™ Super Pulsed Laser MR4™ console (Solon, OH, USA), with the LS50 (emitter with an area of 20 cm2) and SE25 (emitter with an area of 4 cm2) cluster probes as emitters. Nine sites will be irradiated at patient's lumbar region: 3 central sites, using the SE25 (3000 Hz of frequency, 3 minutes of irradiation per site, 24.75 J per site, a totalizing 74.25 J irradiated from SE25); and 6 sites in the same direction, but laterally (both sides, 3 at a side), using the LS50 (1000 Hz of frequency, 3 minutes of irradiation per site, 24.30 J per site, a total of 145.80 J irradiated from LS50). Patients will be treated during 12 sessions over a period of four weeks (three sessions/week). At each treatment session, patients will receive a total dose of 220.05 J. At the end of the 12 treatment sessions, patients will receive a total dose of 2640.60 J.
  Arms: PBMT active

SUMMARY:
Photobiomodulation therapy (PBMT) is a non-pharmacological method commonly used in treatment of musculoskeletal disorders. However, there are few high-quality scientific evidence to support the effectiveness of this therapy in the treatment of patients with chronic low back pain, at short, medium and long term. The present research project aims to evaluate the effects of PBMT in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
This is a randomized, triple-blinded, placebo-controlled trial, with voluntary patients with chronic non-specific low back pain.One hundred and forty-eight patients will be randomly allocated to two treatment groups: Placebo or PBMT for 4 weeks (3 times per week, total of 12 sessions of 27 minutes each). The clinical outcomes will be obtained at the completion of treatment (4 weeks) and at 3, 6 and 12 months after randomization. The data will be collected by a blinded assessor. The statistical analysis will follow the intention-to-treat principles and the between-group differences will be calculated by using mixed linear models.

The outcomes of interest are pain intensity, disability, function and global perceived effect.

ELIGIBILITY:
Inclusion Criteria:

* patients seeking care for chronic non-specific low back pain (defined as pain or discomfort between the costal margins and the inferior gluteal folds, with or without referred symptoms in the lower limbs, for at least 3 month);
* with a pain intensity of at least 3 points measured by a 0-10 points pain numerical rating scale;
* aged between 18 and 65 years;
* able to read Portuguese.

Exclusion Criteria:

* evidence of nerve root compromise (i.e. one or more of motor, reflex or sensation deficit);
* serious spinal pathology (such as fracture, tumor, inflammatory and infectious diseases);
* serious cardiovascular and metabolic diseases;
* previous back surgery;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks after randomization
  Pain intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | 4 weeks after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Pain intensity | 3, 6 and 12 months after randomization
  Pain intensity will be measured by an 11-poin (0-10) Numerical Rating Scale (Pain NRS)
Disability | 3, 6 and 12 months after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire
Function | 4 weeks, 3, 6 and 12 months after randomization
  Function will be measured by an 11-point (0-10) Patient-Specific Functional Scale
Global perceived effect | 4 weeks, 3, 6 and 12 months after randomization
  Global perceived effect will be measured by an 11-point (-5 to +5) Global Perceived Effect Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Oliveira Pena Costa, PhD, Study Director — Universidade Cidade de Sao Paulo
Locations (1):
- Centre for Excellence in Clinical Research in Physiotherapy of Universidade Cidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guimaraes LS, Costa LDCM, Araujo AC, Nascimento DP, Medeiros FC, Avanzi MA, Leal-Junior ECP, Costa LOP, Tomazoni SS. Photobiomodulation therapy is not better than placebo in patients with chronic nonspecific low back pain: a randomised placebo-controlled trial. Pain. 2021 Jun 1;162(6):1612-1620. doi: 10.1097/j.pain.0000000000002189. PMID 33449509
- [Derived] Tomazoni SS, Costa LDCM, Guimaraes LS, Araujo AC, Nascimento DP, Medeiros FC, Avanzi MA, Costa LOP. Effects of photobiomodulation therapy in patients with chronic non-specific low back pain: protocol for a randomised placebo-controlled trial. BMJ Open. 2017 Oct 24;7(10):e017202. doi: 10.1136/bmjopen-2017-017202. PMID 29070637